CLINICAL TRIAL: NCT01319344
Title: Prospective and Open Label Study With Blind End Point Evaluation on the Effect of Mineralocorticoid Receptor Inhibition on Endothelial Function of the Micro- and Macrovasculature in Patients With Metabolic Syndrome
Brief Title: Effect of Eplerenone on Endothelial Function in Metabolic Syndrome
Acronym: MetSyn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MSyn-2010
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Metabolic Syndrome; Endothelial Dysfunction
MeSH Terms: conditions — Metabolic Syndrome | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eplerenone (Experimental)
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 25 mg o.d. per os
  Other Names: Inspra

SUMMARY:
Patients with the metabolic syndrome (MetSyn) are at increased risk for cardiovascular mortality and morbidity.This increased cardiovascular risk is attributed to metabolic dysregulations like impaired glucose tolerance or diabetes mellitus and dyslipidemia, abdominal obesity and arterial hypertension, which promote oxidative stress and inflammation with consecutive endothelial dysfunction causing an atherogenic environment.

Aldosterone promoted end organ damage is mainly found in the cardiovascular system and the kidney. Inflammation and activation of different factors promotes fibroblast growth and matrix production resulting in myocardial fibrosis, vascular remodelling and renal fibrosis.

MetSyn and aldosterone are cardiovascular risk factors and it is of crucial importance to note that there is a connection between MetSyn and aldosterone. Other cross sectional studies show a direct correlation of aldosterone levels and impaired glucose metabolism in patients with and without the MetSyn. Taken together, aldosterone influences essential parameters of the MetSyn. Coincidentally parameters of the MetSyn are stimulus for an increased aldosterone synthesis, i.e. visceral adipocytes.

In large scale clinical trials - RALES, EPHESUS, 4E - inhibition of MR has proven to be beneficial in patients with congestive heart failure and post myocardial infarction and this result has been confirmed for diabetic patients, who are known to have an increased cardiovascular risk.

There is only very limited data on the impact of MR inhibition on metabolic, endocrine, and inflammatory parameters in patients with MetSyn, who have not yet suffered from cardiovascular events.

DETAILED DESCRIPTION:
Patients with the metabolic syndrome (MetSyn) are at increased risk for cardiovascular mortality and morbidity.

This increased cardiovascular risk is attributed to metabolic dysregulations like impaired glucose tolerance or diabetes mellitus and dyslipidemia, abdominal obesity and arterial hypertension, which promote oxidative stress and inflammation and together cause an atherogenic environment. MetSyn is now a well established cardiovascular risk factor and prevalence and incidence of MetSyn in the western world are constantly rising with 19.8 percent prevalence in Germany 4.

Aldosterone is predominantly synthesized in the adrenal glands. In addition, local aldosterone synthesis has been found in the heart and vasculature and aldosterone synthesis in adipocytes is discussed. Aldosterone exerts its effects via the mineralocorticoid receptor (MR). Besides the well described MR in the distal tubule of the kidney MR have also been detected in other organs such as the vasculature and a paracrine mode of action is discussed. Recently it has been described, that MR can be activated independent of aldosterone in hypertensive and obese rats 1. Aldosterone promoted end organ damage is mainly found in the cardiovascular system and the kidney. Inflammation and activation of different factors promotes fibroblast growth and matrix production resulting in myocardial fibrosis, vascular remodelling and renal fibrosis. Aldosterone appears to be involved in all steps of this process by synthesis of reactive oxygen species, induction of inflammation and growth factors like TGF-Beta and connective tissue growth factor. Taken together aldosterone - as the MetSyn- is an independent cardiovascular risk factor 5.

MetSyn and aldosterone are cardiovascular risk factors and it is of crucial importance to note that there is a connection between MetSyn and aldosterone. In clinical studies it was clearly demonstrated that Renin and Aldosterone in patients with MetSyn are elevated 6. Similar results have been obtained in animal studies where obesity induced arterial hypertension increased renin and aldosterone levels 7-9. In a cross sectional study with 397 participants the impact of aldosterone on the onset of arterial hypertension and MetSyn was analysed. In this study blood pressure was associated with aldosterone levels and aldosterone was correlated with waist circumference, insulin, HOMA index and an unfavourable lipid profile 10.

Other cross sectional studies show a direct correlation of aldosterone levels and impaired glucose metabolism in patients with and without the MetSyn 10;11. Taken together, aldosterone influences essential parameters of the MetSyn. Coincidentally parameters of the MetSyn are stimulus for an increased aldosterone synthesis, i.e. visceral adipocytes 12.

In large scale clinical trials - RALES, EPHESUS, 4E 2;3;13 - inhibition of MR has proven to be beneficial in patients with congestive heart failure and post myocardial infarction and this result has been confirmed for diabetic patients, who are known to have an increased cardiovascular risk. In addition, these diabetic patients had significant less hypoglycaemic episodes, indicating an association of MR inhibition and glucose metabolism. Despite the promising data of MR inhibition on cardiovascular mortality and morbidity there is only very limited data on the impact of MR inhibition on metabolic, endocrine, and inflammatory parameters in patients with MetSyn, who have not yet suffered from cardiovascular events.

1. Nagase M, Fujita T. Mineralocorticoid receptor activation in obesity hypertension. Hypertens Res 2009;
2. Pitt B, Reichek N, Willenbrock R et al. Effects of eplerenone, enalapril, and eplerenone/enalapril in patients with essential hypertension and left ventricular hypertrophy: the 4E-left ventricular hypertrophy study. Circulation 2003; 108: 1831-1838
3. Pitt B, Williams G, Remme W et al. The EPHESUS trial: eplerenone in patients with heart failure due to systolic dysfunction complicating acute myocardial infarction. Eplerenone Post-AMI Heart Failure Efficacy and Survival Study. Cardiovasc Drugs Ther 2001; 15: 79-87
4. Moebus S, Hanisch J, Bramlage P et al. Regional Differences in the Prevalence of the Metabolic Syndrome in Primary Care Practices in Germany. Deutsches Ärzteblatt 12, 208-212. 21-3-2008.
5. Milliez P, Girerd X, Plouin PF, Blacher J, Safar ME, Mourad JJ. Evidence for an increased rate of cardiovascular events in patients with primary aldosteronism. J Am Coll Cardiol 2005; 45: 1243-1248
6. Egan BM, Papademetriou V, Wofford M et al. Metabolic syndrome and insulin resistance in the TROPHY sub-study: contrasting views in patients with high-normal blood pressure. Am J Hypertens 2005; 18: 3-12
7. Carroll JF, King JW, Cohen JS. Hydralazine as antihypertensive therapy in obesity-related hypertension. Int J Obes Relat Metab Disord 2004; 28: 384-390
8. Carroll JF, Dwyer TM, Grady AW et al. Hypertension, cardiac hypertrophy, and neurohumoral activity in a new animal model of obesity. Am J Physiol 1996; 271: H373-H378
9. de Paula RB, da Silva AA, Hall JE. Aldosterone antagonism attenuates obesity-induced hypertension and glomerular hyperfiltration. Hypertension 2004; 43: 41-47
10. Kidambi S, Kotchen JM, Grim CE et al. Association of adrenal steroids with hypertension and the metabolic syndrome in blacks. Hypertension 2007; 49: 704-711
11. Goodfriend TL, Egan B, Stepniakowski K, Ball DL. Relationships among plasma aldosterone, high-density lipoprotein cholesterol, and insulin in humans. Hypertension 1995; 25: 30-36
12. Ehrhart-Bornstein M, Arakelyan K, Krug AW, Scherbaum WA, Bornstein SR. Fat cells may be the obesity-hypertension link: human adipogenic factors stimulate aldosterone secretion from adrenocortical cells. Endocr Res 2004; 30: 865-870
13. Pitt D. ACE inhibitor co-therapy in patients with heart failure: rationale for the Randomized Aldactone Evaluation Study (RALES). Eur Heart J 1995; 16 Suppl N: 107-110
14. Grundy SM, Cleeman JI, Merz CN et al. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III Guidelines. J Am Coll Cardiol 2004; 44: 720-732
15. Raff U, Schmidt BMW, Schwab J, Achenbach S, Bär I, Schmieder RE. High incidence of aldosterone breakthrough in therapy resistant hypertension. Journal of Hypertension Suppl. 2009.
16. Schmidt BMW, Raff U, Schwab J, Bär I, Schmieder RE. Eplerenone at low dose induces regression of left ventricular hyprtrophy in resistant hypertension. JASN Suppl. 2008.
17. Schmidt BM, Sammer U, Fleischmann I, Schlaich M, Delles C, Schmieder RE. Rapid nongenomic effects of aldosterone on the renal vasculature in humans. Hypertension 2006; 47: 650-655

ELIGIBILITY:
* Male patients aged > 18 years with mild uncomplicated primary arterial hypertension with a mean sitting SBP ≥ 130 mmHg or DBP ≥ 85 mmHg or treated hypertension and at least 2 of the following traits of the metabolic syndrome (ATP III criteria):

  * abdominal obesity (abdominal girth ≥ 102 cm in males),
  * triglyceride level ≥ 150 mg/dL or treatment for elevated triglyzerides,
  * HDL < 40 mg/dL or treatment for low HDL
  * fasting blood glucose ≥ 100 mg/dL and ≤ 126 mg/dl.
  * Written informed consent
  * Agreement to attend all study visits as planned in the protocol

Exclusion Criteria:

* Patients with or without antihypertensive therapy and mean blood pressure > 160/100 mmHg
* Patients with secondary hypertension
* Patients with one antihypertensive agent maximally dosed or two (or less) agents with half (or less) of maximum approved dose
* Patients with diabetes mellitus type 1 or type 2
* Smokers and ex-smokers < 1 year
* Female patients (to prevent effects of changes in endothelial function attributable to the menstrual cycle)
* Patients with sick sinus syndrome
* Patients with higher degree of sinoatrial or atrioventricular block (II-III)
* Patients with bradycardia (< 50 beats/min)
* Patients with malignant arrhythmias
* Patients with known cardiovascular, disease
* Patients with known cerebrovacular disease
* Patients with peripheral occlusive artery disease
* Patients with history of epilepsy
* Patients with severe hepatic disease (serum GOT, GPT, gamma-GT, AP, bilirubin > 300 of uppper normal range)
* Patients with renal disease defined by eGFR < 60 ml/min/1,73m2
* Patients with history of malignant disease within the last 2 years
* Patients with history of depression
* Patients with drug or alcohol abuse
* Use of any investigational drug within 28 days before study entry
* Known allergy or a known intolerance to the study drug
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol, especially likelihood of the need for additional antihypertensive medication
* Serious disorders which may limit the ability to evaluate the efficacy or safety of the test drug(s), including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematological or oncological, neurological and psychiatric diseases
* Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Subject unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up visits and unlikelihood of completing the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change of basal nitric oxide activity as assessed by change of retinal capillary flow (measured by Scanning Laser Doppler Flowmetry) | Ten weeks

SECONDARY OUTCOMES:
Changes of distensibility of the carotid artery. | Ten weeks
Change of flow mediated dilation of the brachial artery. | Ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof, Principal Investigator — University of Erlangen-Nurnberg
Locations (2):
- Germany (2):
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nurnberg, Erlangen
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Nuremberg

REFERENCES:
- [Derived] Bosch AJ, Harazny JM, Kistner I, Friedrich S, Wojtkiewicz J, Schmieder RE. Retinal capillary rarefaction in patients with untreated mild-moderate hypertension. BMC Cardiovasc Disord. 2017 Dec 21;17(1):300. doi: 10.1186/s12872-017-0732-x. PMID 29268712
- [Derived] Jumar A, Harazny JM, Ott C, Kistner I, Friedrich S, Schmieder RE. Improvement in Retinal Capillary Rarefaction After Valsartan Treatment in Hypertensive Patients. J Clin Hypertens (Greenwich). 2016 Nov;18(11):1112-1118. doi: 10.1111/jch.12851. Epub 2016 Jun 16. PMID 27306560